CLINICAL TRIAL: NCT03960177
Title: An Open-Label, Multi-Institutional Pilot Study to Assess the Use of Glucarpidase in Adult Patients With Osteosarcoma Receiving High-Dose Methotrexate
Brief Title: Glucarpidase After High-Dose Methotrexate in Patients With Osteosarcoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: BTG International Inc. (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Christopher Ryan, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019380; NCI-2019-02257 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00019380 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2019-05-13; First posted 2019-05-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — glucarpidase; gamma-Glutamyl Hydrolase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (glucarpidase) (Experimental): Patients receive standard of care HDMTX IV over 4 hours on day 1 of weeks 4, 5, 9, and 10. After 24 hours after the start of each HDMTX infusion, patients also receive glucarpidase IV over 5 minutes in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Glucarpidase; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Glucarpidase — Given IV
  Other Names: Acetylaspartylglutamate Dipeptidase; Carboxypeptidase G2; carboxypeptidase-G2; CPDG2; CPG2; Poly(gamma-glutamic Acid) Endohydrolase; Pteroylpolygammaglutamyl Hydrolase; Voraxaze
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This early phase I trial studies how well glucarpidase works in reducing toxicity in patients with osteosarcoma receiving high dose methotrexate treatment. Glucarpidase may reduce the levels of methotrexate in patients' blood and lead to shorter hospitalizations and a reduction in toxicities.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rate of completion of 4 planned high dose methotrexate (HDMTX) doses when glucarpidase is administered after each dose.

SECONDARY OBJECTIVES:

I. To assess the length of hospital stay (LOS) associated with methotrexate (MTX) clearance following administration of glucarpidase 24 hours after HDMTX.

II. To assess the LOS associated with all causes following administration of glucarpidase 24 hours after HDMTX.

III. To assess the impact of glucarpidase administration on HDMTX efficacy. IV. To assess the safety and tolerability of 4 doses of HDMTX administered with glucarpidase in an adult osteosarcoma population.

V. To assess the efficacy of glucarpidase flat dose of 1,000 units.

OUTLINE:

Patients receive standard of care HDMTX intravenously (IV) over 4 hours on day 1 of weeks 4, 5, 9, and 10. After 24 and 48 hours after the start of each HDMTX infusion, patients also receive glucarpidase IV over 5 minutes in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up for 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All races and ethnic groups will be eligible

  * A minimum of 6 individuals aged >= 40 years will be enrolled. These participants are considered high-risk.
* Eastern Cooperative Oncology Group (ECOG) performance score 0-2.
* Participants must have pathologically confirmed diagnosis of osteosarcoma. Participants must be newly diagnosed and previously untreated, although initiation of doxorubicin/cisplatin prior to enrollment is permitted.
* Participants must have a recommended treatment plan for their osteosarcoma that includes planned MTX treatment at 8-12 g/m^2.
* Absolute neutrophil count (ANC) >= 1,000/mm^3 (or >= 1.0 x 10^9/L).
* Platelet count 75,000/mm^3 (or >= 75 x 10^9/L).
* Hemoglobin >= 8 g/dL.
* Serum creatinine =< 1.5 x the upper limit of normal (ULN), or glomerular filtration rate (GFR) >= 60 ml/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease (MDRD) formula.
* Total serum bilirubin =< 2 x ULN.
* Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) =< 2.5 x ULN.
* Participants must be willing to use appropriate contraception for the duration of study treatment and four months after completing HDMTX therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Malignant disease, other than those being treated in this study. Exceptions to this exclusion include the following:

  * Malignancies that were treated curatively and have not recurred within 2 years after completion of treatment;
  * Completely resected basal cell and squamous cell skin cancers;
  * Any malignancy considered to be indolent and that has never required therapy;
  * Completely resected carcinoma in situ of any type.
* Participants with rapidly progressive disease or organ dysfunction that would prevent them from receiving planned HDMTX treatment regimen.
* Previous MTX treatment at doses >= 3 g/m^2.
* Previous treatment with glucarpidase.
* Known clinically significant liver disease defined as ongoing drug-induced liver injury, chronic active hepatitis C (HCV), chronic active hepatitis B (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, portal hypertension, or history of autoimmune hepatitis. Patients who have completed curative therapy for HCV are eligible. Patients with known history of human immunodeficiency virus (HIV) infection are eligible.
* Participants with a history of hypersensitivity reactions to study agent or its excipients.
* Participants with a history of hypersensitivity to Escherichia (E.)coli-derived proteins.
* Participants with large pleural or ascitic fluid collection.
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Uncontrolled intercurrent illness, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Unable or unwilling to discontinue use of agents that interact significantly with methotrexate metabolism or excretion.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects completing 4 planned doses of high dose methotrexate (HDMTX) | Time from first dose of HDMTX to time of last dose of HDMTX (week 10)
  Will be estimated with an exact 95% confidence interval (CI).

SECONDARY OUTCOMES:
Length of hospital stay (LOS) for methotrexate (MTX) clearance | Time of start of MTX administration to time of MTX =< 0.1uM sample collection for each planned MTX infusion (up to 15 days)
LOS for all causes (excluding MTX-related AEs) | Date of admission for each planned MTX infusion to date of discharge for each planned MTX infusion (up to 15 days)
Length of hospital stay (LOS) for methotrexate (MTX)-related adverse events (AEs) | Date of admission for each planned MTX infusion to date of discharge for each planned MTX infusion (up to 15 days)
Percent treatment effect at resection | From start of surgery until end of surgery
  Defined as an admixture of degenerating wispy osteoid matrix with empty lacunae, necrotic ghost cells, and edematous stroma with loose fibrous tissue. Dense fibrosis or hyalinization or sheets of sclerotic acellular osteoid may also be present. These features are quantified by estimating the percentage of each parameter in each tumor slide and calculating the mean based on the total number of tumor slides examined. The percentage of tumor necrosis or treatment effect will be recorded from each participant's surgical pathology report.
Incidence of glucarpidase hypersensitivity | From first dose of glucarpidase until 30 days after last dose of glucarpidase
  Will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Will be determined for participants that received at least 1 dose of glucarpidase following an HDMTX infusion. The 95% CI will be reported with the point estimate of toxicity rate.
Incidence of glucarpidase neutralizing antibodies | From first dose of glucarpidase to 30 days after last dose of glucarpidase
  Will be determined for participants that received at least 1 dose of glucarpidase following an HDMTX infusion. The 95% CI will be reported with the point estimate of toxicity rate.
Incidence and severity of MTX-related toxicities | From start of first planned MTX infusion to 30 days after last dose of MTX
  Will be assessed according to CTCAE v 5.0. Will be determined for participants that received at least 1 dose of glucarpidase following an HDMTX infusion. The 95% CI will be reported with the point estimate of toxicity rate.
Incidence and severity of glucarpidase toxicities | From first dose of glucarpidase to 30 days after last dose of glucarpidase
  Will be assessed according to CTCAE v 5.0. Will be determined for participants that received at least 1 dose of glucarpidase following an HDMTX infusion. The 95% CI will be reported with the point estimate of toxicity rate.
MTX and DAMPA serum concentration (umol/L) at 4, 24, 24.5, 36, 48 and every 24 hours after the start of MTX infusion | From start of each planned MTX infusion to time when MTX =< 0.1 uM (for each planned MTX infusion) (up to 15 days)
Proportion of glucarpidase doses (flat dose) that result in MTX serum concentration reduction of >= 97% from hour 24 to hour 24.5 | From first dose of glucarpidase to end of study treatment (week 10)
  Will be presented along with 95% confidence intervals. Summary statistics will be reported on the efficacy analysis set with sub-analyses stratified by glucarpidase dose.
Proportion of glucarpidase doses (flat dose) that result in 48 hour serum MTX level < 1 uM | From first dose of glucarpidase to end of study treatment (week 10)
  Will be presented along with 95% confidence intervals. Summary statistics will be reported on the efficacy analysis set with sub-analyses stratified by glucarpidase dose.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ryan, Principal Investigator — OHSU Knight Cancer Institute
Locations (3):
- United States (3):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - OHSU Knight Cancer Institute, Portland, Oregon
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided